CLINICAL TRIAL: NCT00792883
Title: Clinical Protocol Validation to Identify Prognostic Markers for Critical Care Pediatric Patients
Acronym: PCL07
Status: Completed | Type: Observational
Sponsor: Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, Zina Maria Almeida de Azevedo, PhD, Chief of the pediatric critical care unit of Fernandes Figueira Institute, Oswaldo Cruz Foundation
Other Study IDs: CONEP: 7378
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Sepsis
Keywords: PICU; BIA; Phase angle; RQ; EEM; Compliance; Resistance; Curves; Polymorphisms; NF-kappa B; Scores; PIM 2; PRISM I
MeSH Terms: conditions — Sepsis; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracts from blood or oral swab
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- patients ARDS: 142 Patients in respiratory failure with a diagnosis of ARDS hospitalized at the ICU.
- Patients non ARDS: 432 patients in respiratory failure from other causes (ARDS being formally excluded), hospitalized at the same ICU.
- Healthy controls: 626 healthy patients undergoing elective surgery at the Pediatric Surgery Department or recruited from the pediatric ambulatory.

SUMMARY:
The purpose of this study is to monitor the respiratory, metabolic and nutritional status of critically ill pediatric patients undergoing mechanical ventilation and to correlate the clinical and physiopathological findings with inflammatory activity measurements in order to identify prognostic biomarkers.

DETAILED DESCRIPTION:
Background: Acute Respiratory Distress Syndrome (ARDS) is a frequent cause of respiratory failure in the pediatric intensive care unit (ICU). Bedside respiratory and metabolic monitoring has reduced both morbidity and mortality of children with ARDS in the ICU, and allowed precise evaluation of the gravity of ARDS in individual patients. Recent advances indicate that some ARDS patients present specific, genetically determined profiles of cytokine production, but it is unclear how these relate to systemic inflammation and the gravity of ARDS. It is necessary to define the correlation between genotype, systemic inflammation and prognosis in this group of patients, ir order to define whether they should be targeted for more aggressive anti-inflammatory and immunomodulatory therapy.

Objectives: 1) To evaluate metabolic expenditure,bioelectrical impedance (BIA) and respiratory function in critically ill children undergoing mechanical ventilation. 2) To correlate the metabolic and respiratory parameters with duration of mechanical ventilation, weaning, nutritional status,Phase angle (PA) of BIA, PRISMI and PIM 2 scores in the same children.3) To determine the presence of polymorphisms in the genes for TNF-alfa (- 308 and -863), IL-1ra, IL-6, MIF, LTalfa, il-10 and CD14 in the same children. 4) To define functional parameters of systemic inflammation, including plasma levels of TNF-alfa, IL-1ra, IL-6 and translocation of NF-kappa B in the same children. 5) To correlate genomic and immunological data with PRISM I and PIM 2 scores, PA and mortality.

Methodology: 1) Study Design: A cohort of patients undergoing mechanical ventilation will be submitted to metabolic and respiratory monitoring, and to monitoring of systemic inflammation by measurement of plasma cytokines and NF-kB translocation in peripheral blood leukocytes; a cross-sectional study of cytokine gene polymorphisms will be carried out int hte same population. 2)Subjects: 1000 children, aged 1 mo to 17 yr. Group A: 200 children with ARDS; Group B: 400 children with respiratory failure unrelated to ARDS; Group C (controls): 400 children undergoing preoperatory exams at surgical ward for elective surgery. 3) Methods: Metabolic monitoring: determination of VCO2, VO2, RQ, EEM through indirect calorimetry. Bioelectrical impedance: determination of resistance, reactance and phase angle. Respiratory monitoring: determination of respiratory parameters through capnography, pulse oxymetry, and assessment of respiratory mechanics. Genomic analysis: restriction site mapping and allele-specific amplification by PCR. Immunological evaluation: measurement of plasma cytokines by luminex multiple essays and analysis of NF-kB activation.

ELIGIBILITY:
Inclusion Criteria:

* children aged 1 mo to 17yr undergoing mechanical ventilation in the intensive care unit

Exclusion Criteria:

* chronic inflammatory diseases
* exposure to steroids or other anti-inflammatory agents from anu cause during the month preceding hospitalization.
* malignancies of the immune system (leukemia, lymphoma)

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2007-10; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
mortality | two years

SECONDARY OUTCOMES:
morbidity | two years

CONTACTS AND LOCATIONS:
Overall Officials: Zina Maria A de Azevedo, Principal Investigator — Fernandes Figueira Institute - Fiocruz; Daniella B Moore, Study Chair — Fernandes Figueira Institute - Fiocruz
Locations (1):
- Instituto Fernandes Figueira, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Azevedo ZM, Moore DB, Lima FC, Cardoso CC, Bougleux R, Matos GI, Luz RA, Xavier-Elsas P, Sampaio EP, Gaspar-Elsas MI, Moraes MO. Tumor necrosis factor (TNF) and lymphotoxin-alpha (LTA) single nucleotide polymorphisms: importance in ARDS in septic pediatric critically ill patients. Hum Immunol. 2012 Jun;73(6):661-7. doi: 10.1016/j.humimm.2012.03.007. Epub 2012 Apr 13. PMID 22507624